CLINICAL TRIAL: NCT06661434
Title: Prevalence of Obesity Among Adult Patients With Congenital Heart Disease: a Population-based Study
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Annette Schophuus Jensen, MD PhD, Rigshospitalet, Denmark
Other Study IDs: R-21066074
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Congenital Heart Disease
Keywords: obesity; adult congenital heart disease
MeSH Terms: conditions — Obesity; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study was conductede to examined the prevalence of obesity in a large Danish ACHD cohort, stratified according to age, sex and disease severities. To do so, ACHD patients were matched by age and sex with controls from the contemporary Copenhagen General Population Study

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart disease
* BMI within the last five years

Exclusion Criteria:

* Without BMI or not congenital heart disease

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The ACHD population in east Denmark
Sampling Method: Non-Probability Sample
Enrollment: 7157 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
BMI | Within the last five years
  Body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No